CLINICAL TRIAL: NCT03647579
Title: Effect of Single Dose Dexmedetomidine Versus Midazolam on Emergence Agitation and Recovery Profile When Added to Ketamine for Procedural Sedation and Analgesia in Pediatric Patients Undergoing Bone Marrow Aspiration and Biopsy
Brief Title: Dexmedetomidine Versus Midazolam Added to Ketamine in Pediatric Patients Undergoing Bone Marrow Aspiration and Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed H Othman, Assisstant professor of Anesthesia ICU and pain Relief, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17100208
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Procedural Sedation and Analgesia During Bone Marrow Aspiration and Biopsy
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- midazolam plus ketamine (Active Comparator)
  Interventions: Drug: midazolam intravenous infusion of 0.05 mg/kg plus 1 mg/kg ketamine
- dexmedetomidine plus ketamine (Active Comparator)
  Interventions: Drug: Dexmedetomidine intravenous infusion of 2mic/kg plus 1 mg/kg ketamine

INTERVENTIONS:
Drug: midazolam intravenous infusion of 0.05 mg/kg plus 1 mg/kg ketamine — midazolam intravenously (i.v.) in a dose of 0.05 mg/kg diluted by 50ml saline over 10 minutes using syringe pump plus 1 mg/kg ketamine
  Arms: midazolam plus ketamine
Drug: Dexmedetomidine intravenous infusion of 2mic/kg plus 1 mg/kg ketamine — Dexmedetomidine intravenously (i.v.) in a dose of 2mic/kg diluted by 50ml saline over 10 minutes using syringe pump plus 1 mg/kg ketamine
  Arms: dexmedetomidine plus ketamine

SUMMARY:
Group I :The patients will receive midazolam intravenously (i.v.) in a dose of 0.05 mg/kg diluted by 50ml saline over 10 minutes using syringe pump plus 1 mg/kg ketamine (iv).

Group II : The patients will receive Dexmedetomidine intravenously (i.v.) in a dose of 2mic/kg diluted by 50ml saline over 10 minutes using syringe pump plus 1 mg/kg ketamine (iv).

The objective of this study to evaluate the clinical effects, adverse effects and recovery time of two different sedative agents (midazolam and Dexmedetomidine) combined with ketamine during conscious sedation for child patient with haematological cancer undergoing BMA &biopsy.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive children with acute lymphoblastic leukemia undergoing bone marrow aspiration and biopsy.

Exclusion criteria:

* previous sensitization or anaphylactic reaction to Dexmedetomidine, ketamine,and midazolam;
* evidence of head injury,
* raised intracranial or intraocular tension;
* use of drugs known to interact with either study agent;
* an American Society of Anesthesiologists (ASA) physical status score greater than 2.
* Also Patients with cardiovascular, respiratory, hepatic diseases and epilepsy will be excluded.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
efficacy of drug mixture on procedural sedation and analgesia: Ramsay sedation score | within the time of the procedure of bone marrow aspirate and biopsy
  to assess efficacy of procedural sedation and analgesia with drug mixture;using Ramsay sedation score.
  Ramsay score
  1. Nervous, agitated, and/or restless.
  2. Cooperative, orientated, quite patient.
  3. Only obeying orders.
  4. Sleeping, hitting the glabella, and responding to high voice suddenly
  5. Sleeping, hitting the glabella, and responding to high voice slowly
  6. No response to any of these stimulations Dexemeditomidine and midazolam will be started 2 minutes before procedure through a peripheral venous cannula and continued as maintainance, then ketamine will be administered over 10-20 s aiming to achieve a sedation level of 3 or 4 on Ramsay scale to start the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Institute, Assiut University, Asyut, Egypt